CLINICAL TRIAL: NCT01710826
Title: A Single-center, Double-blind, Randomized, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ascending 14-day Repeated Oral Doses of Genz-682452 in Healthy Male and Female Subjects
Brief Title: A Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Genz-682452 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GZFD00311; TDR12768 (Other: Sanofi)
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
MeSH Terms: interventions — venglustat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genz-682452 (Experimental): This study will include three cohorts for doses of Genz-682452: Dose 1, Dose 2, Dose 3. Each cohort will include 12 participants, 9 of whom will be administered Genz-682452 and 3 will be administered placebo.
  Interventions: Biological: Genz-682452
- Placebo (Placebo Comparator): Placebo comparator taken by participants randomized to the placebo arm in each of the three cohorts. Each cohort will include 12 participants, 9 of whom will be administered Genz-682452 and 3 will be administered placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Genz-682452 — Capsules for oral administration.
  Arms: Genz-682452
Biological: Placebo — Placebo capsules matching the Genz-682452 capsules.
  Arms: Placebo

SUMMARY:
To assess in healthy adult subjects:

* The tolerability and safety of ascending repeated oral doses of Genz-682452.
* The pharmacokinetic parameters of Genz-682452 after ascending repeated oral doses.
* The pharmacodynamics of Genz-682452 after ascending repeated oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50.0 and 95.0 kg, inclusive, if male and between 40.0 and 85.0 kg inclusive, if female, body mass index between 18.0 and 30.0 kg/m^2, inclusive.
* Certified as healthy by a comprehensive clinical assessment.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting.
* Blood donation, any volume, within 2 months before inclusion.
* Symptomatic postural hypotension.
* History or presence of drug or alcohol abuse.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, antihepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Participants with Treatment-Emergent Adverse Events (TEAEs) | Day 1 through Day 14

SECONDARY OUTCOMES:
Pharmacokinetics as measure by plasma parameters | Day 1 through Day 14
  Maximum plasma concentration (Cmax), Plasma Concentration Observed Just Before Treatment Administration During Repeated Dosing (Ctrough), First time to reach Cmax (Tmax), Area Under the Plasma Concentration Versus Time Curve Over the Dosing Interval 0-23 hours (AUC0-24), Terminal Half-Life (t1/2z), Apparent Total Body Clearance of Genz-682452 at steady state (CLss/F), plasma 4 beta-hydroxycholesterol (4β-HC)
Pharmacodynamics as measure by Plasma concentrations of Glucosylceramide (GL-1), Globotriaosylceramide (GL-3) and GM3 ganglioside (GM3) | Day 1, through Day 14
Pharmacokinetics Urine parameter as measure by assessment of Genz-682452 in Urine, Ae0-t, fe0-t (Exploratory) | Day 1 through Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Austin, Texas, United States

REFERENCES:
- [Derived] Peterschmitt MJ, Crawford NPS, Gaemers SJM, Ji AJ, Sharma J, Pham TT. Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Oral Venglustat in Healthy Volunteers. Clin Pharmacol Drug Dev. 2021 Jan;10(1):86-98. doi: 10.1002/cpdd.865. Epub 2020 Aug 26. PMID 32851809